CLINICAL TRIAL: NCT06575231
Title: Accuracy and User Performance Evaluation of PixoTest HbA1c Measurement System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CMUH105-REC1-080
Record Dates: First submitted 2024-08-22; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Diabetes; HbA1c
Keywords: HbA1c
MeSH Terms: conditions — Diabetes Mellitus | interventions — In Vitro Meat

STUDY DESIGN:
Intervention Model Description: Each subject should draw two tubes of venous blood in the K2-EDTA. One tube should be tested by POC operator as a study participant using the PixoTest POCT System. The other tube takes 1c.c. blood sample from K2-EDTA to analyzed with a comparison method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Type 2 diabetic patients (Experimental): 1. 20 years or older.
  2. Willing to participate in the study, able to read and provide written informed consent form.
  3. HCT 25~65%.
  4. Subjects including healthy subjects, outpatients, and inpatients.
  Interventions: Diagnostic Test: in-vitro

INTERVENTIONS:
Diagnostic Test: in-vitro — responding smartphone. It is intended for quantitative measurement of HbA1c in capillary whole blood and use in the home by people with diabetes mellitus as an aid to monitor the effectiveness of diabetes control.

SUMMARY:
To evaluate the accuracy user performance of PixoTest HbAc1 measurement system and to collect feedback from subjects.

DETAILED DESCRIPTION:
According to WHO report, the number of people with diabetes has risen from 108 million in 1980 to 422 million in 2014. Diabetes is a major cause of blindness, kidney failure, heart attacks, stroke and lower limb amputation. In 2012 alone diabetes caused 1.5 million death. Tight glucose control is essential for prevention of complications in people with diabetes. The Diabetes Control and Complications Trial (DCCT) provided direct evidence the relationship between HbA1c level and risks for diabetic complications in diabetes. Based on the results of the DCCT, the American Diabetes Association (ADA) has published recommendations for HbA1c and plasma glucose levels that are widely used. HbA1c testing can be performed at any time of day and without special patient preparation, it is more convenient for patients and even measuring fasting plasma glucose.

The ADA recommends measurement of HbA1c (typically 3-4 times per year for type 1 and poorly controlled type 2 diabetic patients, and 2 times per year for well-controlled type 2 diabetic patients) to determine whether a patient's metabolic control has remained continuously within the target range. .Most diabetes patients will go to hospital to measurement HbA1c, but should wait few days for test result. Most diabetes patient maybe not measurement HbA1c so many time per year. The PixoTest HbA1c measurement system can give result for a few minutes at home. The diabetes patient can measure HbA1c at home don't need go to hospital.

The PixoTest HbA1c measurement system is defined as the respective reagent system and the corresponding smartphone. It is intended for quantitative measurement of HbA1c in capillary whole blood and use in the home by people with diabetes mellitus as an aid to monitor the effectiveness of diabetes control.

This study is designed to test the accuracy and user performance of the Pixotest HbA1c measurement system.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older.
2. Willing to participate in the study, able to read and provide written informed consent form.
3. HCT 25~65%.
4. Subjects including healthy subjects, outpatients and inpatients.

Exclusion Criteria:

1. An individual who does not meet the inclusion criteria will be excluded from enrollment.Taking prescription anticoagulants (such as Warfarin or Heparin) or have clotting problems that may prolong bleeding. Taking Plavix or aspirin daily is not excluded.
2. Hemophilia or any other bleeding disorder
3. Reports having an infection with a blood borne pathogen (e.g. HIV, hepatitis)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-05-17 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
HbA1c | 3 minutes
  HbA1c testing can be performed at any time of day and without special patient preparation.

CONTACTS AND LOCATIONS:
Overall Officials: Shi-Yann Cheng, M.D, Principal Investigator — China Medical University Beigang Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NGSP Manufacturer Certified Methods — https://ngsp.org/index.asp